CLINICAL TRIAL: NCT07193186
Title: A Phase II Study of Anlotinib and Benmelstobart as Second-line Treatment in Locally Advanced or Metastatic Differentiated Thyroid Cancer
Brief Title: Anlotinib and Benmelstobart in DTC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Yu Wang, Chief of Head and Neck Surgery, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABILITY
Record Dates: First submitted 2025-09-18; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms | interventions — anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Benmelstobart+Anlotinib
  Interventions: Drug: Anlotinib and Benmelstobart

INTERVENTIONS:
Drug: Anlotinib and Benmelstobart — Patients will receive Benmelstobart (1200mg, d1, q3w) in combination with Anlotinib (12mg, qd, d1-14, q3w). Treatment will continue until disease progression, voluntary withdrawal of informed consent, intolerable toxicity, or until the investigator determines that the patient no longer benefits.

SUMMARY:
This study is a multicenter, open-label, phase II study to evaluate the efficacy and safety of Benmelstobart in combination with Anlotinib as a second-line treatment for locally advanced or metastatic differentiated thyroid cancer. Patients who meet the inclusion criteria and do not meet the exclusion criteria will receive Benmelstobart (1200mg, d1, q3w) in combination with Anlotinib (12mg, qd, d1-14, q3w). Treatment will continue until disease progression, voluntary withdrawal of informed consent, intolerable toxicity, or until the investigator determines that the patient no longer benefits. For locally advanced patients, if the disease converts from unresectable or borderline unresectable to resectable after treatment, surgical intervention will be performed.

ELIGIBILITY:
Inclusion Criteria:

* The patient voluntarily agrees to participate in this study and has signed the informed consent form;
* Age: ≥18 years, regardless of gender;
* Histologically confirmed differentiated thyroid cancer;
* Unresectable or borderline unresectable locally advanced thyroid cancer and/or metastatic thyroid adenocarcinoma;
* Failure of first-line treatment (failure to achieve partial or complete response) or disease progression after first-line treatment;
* At least one measurable lesion;
* ECOG PS: 0-2;
* Expected survival period ≥12 weeks;
* Patient agrees to undergo tumor tissue biopsy/surgery at the time of enrollment;
* Normal function of major organs;
* Willingness to use reliable contraceptive methods during the trial. Women of childbearing potential must have a negative pregnancy test (serum or urine) within 14 days prior to enrollment.
* The subject voluntarily agrees to participate in this study, signs the informed consent form, demonstrates good compliance, and cooperates with follow-up.

Exclusion Criteria:

* Presence of other active malignancies within the past 5 years or concurrently. Patients with cured localized tumors, such as basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, carcinoma in situ of the prostate, carcinoma in situ of the cervix, carcinoma in situ of the breast, etc., may be enrolled.
* Use of other antitumor therapies (including but not limited to chemotherapy, radiotherapy, etc.) within 28 days prior to the first administration of the study drug. Thyrotropin (TSH) suppressive therapy is excluded.
* Prior treatment with immune checkpoint inhibitors (including but not limited to nivolumab, pembrolizumab, toripalimab, sintilimab, etc.).
* Any severe or uncontrolled systemic disease, as determined by the investigator, including poorly controlled hypertension (systolic blood pressure >160 mmHg or diastolic blood pressure >100 mmHg) despite medication, uncontrolled diabetes, poorly managed cardiac disease, and signs of active bleeding.
* Known history of severe allergy to any monoclonal antibody or anti-angiogenic targeted drug.
* Presence of uncontrolled infection at the time of screening.
* Pregnant or lactating women.
* Refusal to undergo tumor tissue biopsy at the time of enrollment.
* Other conditions considered by the treating physician as unsuitable for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate，ORR | 2 years
  Objective Response Rate (ORR) as assessed based on RECIST 1.1 criteria.

IPD SHARING:
Plan to Share IPD: Undecided